CLINICAL TRIAL: NCT05141916
Title: Optimizing the Evaluation and Management of Patients With Suspected Choledocholithiasis
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB18-1053
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Biliary Disease; Choledocholithiasis
MeSH Terms: conditions — Gallbladder Diseases; Choledocholithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholagiopancreatography (ERCP) — Endoscopic procedure employed to manage biliary and pancreatic diseases

SUMMARY:
Choledocholithiasis (stone(s) in the common bile duct) is common. Untreated or missed, choledocholithiasis has high morbidity and mortality. Endoscopic retrograde cholangio-pancreatography (ERCP) is recognized as the first-line modality for management. While effective, ERCP is associated with adverse events. Thus, the selection of patients for ERCP should be accompanied by a high pre-test suspicion of choledocholithiasis.

Choledocholithiasis is suspected based on clinical, biochemical and radiographic findings. The most relied-upon strategy for risk stratification of choledocholithiasis is based on guidelines from The American Society for Gastrointestinal Endoscopy (ASGE). In it, clinical predictors are defined as "very strong", "strong" or "moderate", and the presence of one or more of these is meant to suggest "high" or "intermediate" probability of choledocholithiasis.

A knowledge gap exists in the performance characteristics of intermediate-probability criteria, where overall accuracy is <50% from limited data. Patients in this group are recommended to a) undergo endoscopic ultrasound (EUS) or magnetic resonance cholangio-pancreatography (MRCP), b) undergo cholecystectomy with intra-operative cholangiography (IOC), or c) proceed directly to ERCP. At centres where EUS and MRCP are readily available, these are preferred options, as they are least invasive and sensitive; however, they are often unavailable. Thus, in clinical practice, a high proportion of intermediate-risk patients ultimately proceed directly to ERCP, where likelihood of benefit is only moderate, while procedural risk remains.

The role of liver enzyme changes has not been evaluated; however, dynamic changes may offer another method for evaluating patients at intermediate risk of CBD stones that is safe and available. Incorporation of dynamic liver enzymes may improve the test-performance characteristics of the existing framework.

DETAILED DESCRIPTION:
There are two planned phases for this proposed study. The first will be a retrospective phase aimed at assessing the test performance characteristics of the current guideline-based criteria, and subsequently with developing a novel with the incorporation of dynamic liver enzyme changes into the intermediate-probability CBD stone management algorithm. In the second phase, we will evaluate and prospectively validate the proposed model.

Phase 1 - Retrospective Evaluation

This will be a retrospective study of patients evaluated for suspected choledocholithiasis. Given the nature of our tertiary care facility as outlined above, this will constitute a population-based study of a sample of 1,000 patients from 2012-2017 who underwent evaluation for choledocholithiasis. The selection of 2012 as the start of our study period is based on an appropriate time lag from publication to widespread clinical adoption of the ASGE guidelines, which were published in 2010.

An institutional endoscopy database and reporting platform (Endopro, Pentax) has been used in Calgary since 2000, and it is estimated that well over 95% of all ERCP and EUS procedures have been reported using Endopro since its implementation. We will employ several strategies to capture patients. We will initially search our Endopro database for all ERCPs and EUS exams performed where the indication was "suspected choledocholithiasis" of any probability. This broad search strategy will identify all possible choledocholithiasis cases. Potential cases will then be grouped by patient name and ordered by data.

Once the potential cases are gathered, and the appropriate sample of 1,000 extracted, a manual review of each of the endoscopy reports will be performed, in addition to a review of the patients' medical records through Sunrise Clinical Manager, by one of two independent medical reviewers.

Patient baseline demographics (age, gender), co-morbidities and medications will be recorded. In addition, available laboratory parameters will be recorded for the 7 days preceding the procedure, allowing for the assessment of trends. Any relevant diagnostic imaging tests performed in the preceding 60 days will also be captured.

A positive diagnosis of choledocholithiasis will be defined as the presence of stone(s), sludge, debris or microlithiasis on a definitive study (ERCP or IOC). Where our proposed study will differ from previous studies with similar designs is that we will also incorporate a follow-up period, where a negative diagnosis of choledocholithiasis will require that a patient has no readmissions, repeat visits or medical procedures related to choledocholithiasis within 6 months of the initial period of clinical suspicion.

Using the above extracted data, we will be able to determine the performance characteristics of relevant parameters in the evaluation of choledocholithiasis, in addition to assessing the utility of dynamic enzyme trends. New framework(s) and/or novel criteria will then be developed using the findings, that select the optimal blend of test characteristics both for ruling in and ruling out choledocholithiasis.

Phase 2 - Prospective Validation

The novel algorithm developed in Phase 1 will then be applied in a prospective fashion, when possible, to consecutive patients undergoing EUS or ERCP for suspected choledocholithiasis. The same variables will be measured as in Phase 1, but in Phase 2, a research assistant (RA) will prospectively enter data and follow up with patients. The sequence of procedures will be as follows:

1. The patient is referred to PLC Endoscopy Unit for consideration of ERCP or EUS procedure, and is booked by the attending advanced/therapeutic endoscopist on call as appropriate, as per the standard of care.
2. All patients referred to this service are either a) outpatients or b) inpatients.

   1. Outpatients will be ineligible for the study as per our defined exclusion criteria in Section 3.3.
   2. Inpatients, once verbal and written consent to approach has been given to their admitting nurse, will be approached by the RA prior to their procedure to discuss the actively enrolling study, and to answer any potential questions. Inpatients with suspected or proven cholangitis will be excluded since it is generally agreed that these patients should proceed directly to ERCP.
3. If the patient agrees to participate, the relevant informed database/study consent form(s) is/are signed and witnessed. If the patient decides not to participate, the ERCP or EUS proceeds as per the usual standard of care (and the sequence that follows does not apply).
4. The RA collects any relevant patient-related and pre-procedural data through combination of direct patient interview and subsequent review of the medical records.
5. The patient is then met by the endoscopist performing the procedure to discuss the risks and benefits of the procedure and have the patient sign informed consent for the procedure.The patient enters the endoscopy/fluoroscopy room and the procedure commences.
6. During the procedure, relevant peri-procedural data are recorded by the RA by direct observation, and/or, if necessary, in consultation with the procedural physician(s) and/or nurse(s).
7. After the procedure is complete, the patient is moved to the recovery room for observation. Depending on their disposition and the course of the procedure, observation times and protocols differ. During this stage, the RA collects any relevant post-procedural data, and any missing pre- or peri-procedural data.
8. Any peri- or immediate post-procedural adverse event is recorded prospectively in the database.
9. The patient is examined by the endoscopist prior to discharge and provided with written post-procedure information, including a phone number to call in the event of any issues.
10. The RA meets with the patient prior to their discharge from the unit to answer any final potential questions.
11. Any formal histology or cytopathology results from the procedure are recorded in the database by the RA as they become available.
12. Patients are contacted by the RA by telephone 30 days following their procedure to assess ongoing symptoms and advise of any adverse events, including emergency department visits or inpatient admissions. If any are endorsed, the details are captured electronically.
13. The patient medical record is reviewed 6 months following their procedure to assess for any adverse events, including emergency department visits, inpatient admissions, repeat procedures or surgeries related to a possible diagnosis of choledocholithiasis. The details are captured electronically.
14. Any potential study outcomes will then be analyzed and presented in manuscript form, and submitted to peer reviewed journals for eventual publication as well as to conferences for dissemination.
15. All participants will be mailed a letter outlining the results of any relevant studies, and thanking them for their involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected choledocholithiasis, regardless of probability
* age 18 years old or older
* able to give informed consent to involvement (in the prospective validation phase).

Exclusion Criteria:

* Unable or unwilling to provide informed consent;
* age < 18 years;
* suspected or proven cholangitis;
* previous ERCP with sphincterotomy;
* prior diagnosis or management of choledocholithiasis;
* outpatient status;
* out-of-province status (prohibiting full medical record access).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing ERCP for suspected choledocholithiasis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Positive or negative diagnosis of choledocholithiasis | immediate
  Retrospective analysis will be employed to determine the individual and joint test performance characteristics of the parameters in the ASGE guideline, and to determine the (lone and additional) test characteristics of dynamic enzyme changes, in predicting the primary outcome measure. The agreed-upon model will then be validated prospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Nauzer Forbes, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-specific data will be in a de-identified encrypted secure format whenever shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: For 5 years after data collection is complete.
Access Criteria: Deidentified aggregate level data can be shared upon reasonable request.